CLINICAL TRIAL: NCT02066337
Title: Effect of Ozone Gel on Alveolar Bone Density and Superoxide Dismutase in Chronic Periodontitis: A Randomized Controlled Clinical Study
Brief Title: Effect of Ozone Gel on Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Lecuture, October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mn1965
Record Dates: First submitted 2014-01-30; First posted 2014-02-19 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Periodontal Diseases
Keywords: Ozone gel; Antioxidants; Chronic periodontitis; Superoxide dismutase
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo gel (Placebo Comparator): scaling and root planing with placebo gel
  Interventions: Procedure: scaling and root planing; Drug: placebo gel
- Ozonated olive oil gel (Active Comparator): scaling and root planing with Ozonated olive oil gel
  Interventions: Procedure: scaling and root planing; Drug: Ozonated olive oil gel

INTERVENTIONS:
Procedure: scaling and root planing
Drug: placebo gel
  Arms: placebo gel
Drug: Ozonated olive oil gel
  Other Names: Ozonated olive oil gel = Oxactiv gel
  Arms: Ozonated olive oil gel

SUMMARY:
To evaluate the efficacy of locally delivered ozone gel as an adjunct to conventional periodontal therapy on selected clinical parameters as well as alveolar bone density (BD) and superoxide dismutase (SOD) activity in patient with chronic periodontitis.

DETAILED DESCRIPTION:
In this study, the investigators tested the effect of ozone gel as a local delivery system in treatment of chronic periodontitis in term of probing pocket depth reduction, mean gain in clinical attachment level, a more rise in BD values as well as greater reduction in SOD activity compared to scaling and root planing (SRP) alone.

ELIGIBILITY:
Inclusion Criteria:

1. The participant's age ranged between 30 and 60 years.
2. All of the patients suffered from chronic periodontitis with attachment loss ≥ 5mm.
3. Willingness to participate and sign the informed consent.

Exclusion Criteria:

1. Any systemic disease that affect the periodontium.
2. Pregnancy, lactation, postmenopausal women
3. People who take anti-inflammatory drugs, antibiotics or vitamins within the previous 3 month.
4. People who use mouth washes regularly
5. Heavy smoking (> 10 cigarettes/day)
6. History of alcohol abuse.
7. Participation in other clinical trials.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Superoxide dismutase activity | 6 months
  Superoxide dismutase activity in the gingival crevicular fluid was carried out at baseline, 1, 3 and 6 months post treatment.

SECONDARY OUTCOMES:
Plaque Index | 6 months
  plaque index was recorded at baseline and at 1, 3 and 6 months post treatment.
Gingival index | 6 months
  Gingival index was recorded at base line,1,3,6 months post treatment
Probing pocket depth | 6 months
  Probing pocket depth was recorded at base line, 1, 3, 6 months post treatment
Clinical attachment level | 6 months
  Clinical attachment level was recorded at baseline, 1, 3 and 6 months post treatment
Bone density | 6 months
  Bone density was carried out using Digora software (Digora system, Soredex, Orion Corp., Finland) at baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Enas Elgendy, ph.D, Principal Investigator — October 6 University
Locations (1):
- October 6 University, Cairo, Egypt